CLINICAL TRIAL: NCT01867385
Title: The Physiology of Fatigue in Patients With Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130142; 13-DK-0142
Record Dates: First submitted 2013-05-31; First posted 2013-06-04 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11-20

CONDITIONS: Liver Disease
Keywords: Fatigue; Chronic Hepatitis; Chronic Hepatitis B; Chronic Hepatitis C; Hepatitis
MeSH Terms: conditions — Liver Diseases; Fatigue; Hepatitis, Chronic; Hepatitis B, Chronic; Hepatitis C, Chronic; Hepatitis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Fatigue is a common and often disabling symptom in people with chronic liver disease. Its causes are not well understood. Sleep disturbance may play a role in people with cirrhosis, but these factors have not been studied in people with other stages of liver disease. This study will look at the body's circadian rhythms (internal clock) to see if problems with these rhythms can contribute to fatigue. It will look at the causes and mechanisms of fatigue in people with chronic liver disease by comparing people with and without fatigue.

Objectives:

- To study reasons for fatigue in people with chronic liver disease.

Eligibility:

* <TAB>Individuals at least 18 years of age who have chronic liver disease.
* <TAB>Participants with or without fatigue may enroll.

Design:

* Participants will be screened with a physical exam and medical history. They will have a 2-day inpatient stay for the study.
* For the 7 days before the inpatient stay, participants will keep a sleep diary. They will record any caffeine or alcohol consumption, medicines, exercise, and sleep or naps. They will also wear an actigraph to measure their activity levels.
* During the inpatient stay, participants will answer questions about fatigue and sleep habits. They will have regular blood tests for 24 hours. Their body temperature will also be monitored. During the night, they will have a sleep study to look at how well or poorly they sleep.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Fatigue is a common symptom in patients with chronic liver disease, and can severely impact quality of life. Thus far, there is scant knowledge about the causes of fatigue in this population, and almost no specific treatments for fatigue have been found effective in clinical trials. Sleep disturbance and alterations in plasma melatonin profiles have been documented in patients with cirrhosis, but remain largely unstudied in patients with earlier stages of liver disease. Up to 50 patients will be enrolled in a case-control study on the physiology of fatigue in patients with chronic liver disease. This is a descriptive study, exploring the concept that fatigue may be the result of circadian rhythms in the central nervous system being out of sync with circadian rhythms in peripheral organs, i.e. unsynchronized central and peripheral clocks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults (age >18) with chronic liver disease of any etiology

EXCLUSION CRITERIA:

* Treatment with medications or supplements frequently associated with fatigue, such as interferon (within the last four months), beta-blockers, calcium channel blockers, benzodiazepines, sedating antihistamines, antidepressants, antipsychotics, or melatonin. In select instances, patients using these medications may be enrolled if, in the opinion of the investigators, their fatigue is clearly unrelated to the medication.
* Untreated or uncontrolled comorbidities that influence fatigue, including thyroid disorders (TSH>5 mcIU/mL), anemia (Hemoglobin<11 g/dL), major depression, active substance abuse or other conditions as determined by the enrolling physician. Comorbidities that are adequately controlled will not exclude patients.
* Untreated sleep disorders such as obstructive sleep apnea or restless leg syndrome
* Decompensated cirrhosis (encephalopathy, gastrointestinal bleeding, ascites, bilirubin >2) within the last six months
* Patients planning to travel outside the time zone during the study period
* Known or suspected significant gastrointestinal motility disorder, obstruction, or structuring disease
* Pregnancy, breastfeeding, or intention to become pregnant
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05-31; Primary Completion 2015-09-11 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Circadian rythms | 2-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Foster GR, Goldin RD, Thomas HC. Chronic hepatitis C virus infection causes a significant reduction in quality of life in the absence of cirrhosis. Hepatology. 1998 Jan;27(1):209-12. doi: 10.1002/hep.510270132. PMID 9425939
- [Background] Gumber SC, Chopra S. Hepatitis C: a multifaceted disease. Review of extrahepatic manifestations. Ann Intern Med. 1995 Oct 15;123(8):615-20. doi: 10.7326/0003-4819-123-8-199510150-00008. PMID 7677303
- [Background] Kallman J, O'Neil MM, Larive B, Boparai N, Calabrese L, Younossi ZM. Fatigue and health-related quality of life (HRQL) in chronic hepatitis C virus infection. Dig Dis Sci. 2007 Oct;52(10):2531-9. doi: 10.1007/s10620-006-9708-x. Epub 2007 Apr 4. PMID 17406828